CLINICAL TRIAL: NCT07129382
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase Ib/II Study to Evaluate the Efficacy and Safety of CS32582 Capsule in Adult Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of CS32582 in Participants With Moderate to Severe Plaque Psoriasis
Acronym: MECAP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS32582-201
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1：Low dose CS32582 (Experimental): The patient received low-dose CS32582 capsules BID or placebo for 4 weeks
  Interventions: Drug: CS32582 capsule（low dose） or matched placebo
- Part 1：Hgh dose CS32582 (Experimental): The patient received high-dose CS32582 capsules BID or placebo for 4 weeks
  Interventions: Drug: CS32582 capsule（high dose） or matched placebo
- Part 2：Low dose CS32582 (Experimental): The patient received low-dose CS32582 capsules BID or placebo for 12 weeks
  Interventions: Drug: CS32582 capsule（low dose）
- Part 2：Medium dose CS32582 (Experimental): The patient received medium-dose CS32582 capsules BID or placebo for 12 weeks
  Interventions: Drug: CS32582 capsule（medium dose）
- Part 2：High dose CS32582 (Experimental): The patient received high-dose CS32582 capsules BID or placebo for 12 weeks
  Interventions: Drug: CS32582 capsule（high dose）

INTERVENTIONS:
Drug: CS32582 capsule（low dose） or matched placebo — CS32582 capsule（low dose） or matched placebo，4 weeks
  Arms: Part 1：Low dose CS32582
Drug: CS32582 capsule（high dose） or matched placebo — CS32582 capsule（high dose） or matched placebo，4 weeks
  Arms: Part 1：Hgh dose CS32582
Drug: CS32582 capsule（low dose） — CS32582 capsule（low dose），12 weeks
  Arms: Part 2：Low dose CS32582
Drug: CS32582 capsule（medium dose） — CS32582 capsule（medium dose），12 weeks
  Arms: Part 2：Medium dose CS32582
Drug: CS32582 capsule（high dose） — CS32582 capsule（high dose），12 weeks
  Arms: Part 2：High dose CS32582

SUMMARY:
" This study consists of two parts: Part 1 (Dose Escalation): A randomized, double-blind, placebo-controlled phase in which approximately 20 to 30 adult patients with plaque psoriasis will receive the investigational treatment for 4 weeks.

Part 2 (Efficacy and Safety Assessment): A randomized, double-blind, placebo-controlled evaluation where approximately 200 adult patients with plaque psoriasis will undergo 12 weeks of treatment.

The resulting data will provide preliminary evidence on the safety and efficacy profile of CS32582, informing its subsequent development strategy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form (ICF) after fully understanding the trial.
* Age 18-70 years (inclusive) at consent, any gender
* Clinically diagnosed with chronic plaque psoriasis, defined as disease duration ≥ 6 months at screening.
* Stable plaque psoriasis at screening, defined as no significant flare-ups or morphological changes during the 6 months prior to screening (investigator-assessed).
* Moderate-to-severe disease at screening/randomization: PASI≥12, sPGA≥3, and BSA≥10%;
* Candidate for phototherapy or systemic therapy per investigator's judgment.
* Women of childbearing potential and males: Agreement to use highly effective contraception from consent until 30 days post-last dose.

Exclusion Criteria:

* Forms of psoriasis other than plaque-type (e.g., erythrodermic, pustular, guttate, or drug-induced psoriasis) .
* Presence of other skin conditions that in the judgement of the Investigator could interfere with study assessment.
* Immune-mediated diseases requiring systemic therapy (e.g., inflammatory bowel disease), except NSAIDs.
* History of severe drug allergies.
* Major surgery within 2 months before randomization or planned during the study.
* Drug/alcohol abuse within 6 months before screening.
* Uncontrolled hypertension at screening (SBP >160 mmHg or DBP >100 mmHg).
* Myocardial infarction, unstable angina, TIA, stroke, PCI, or CABG within 6 months before screening.
* NYHA Class III/IV heart failure at screening.
* History of malignancy or lymphoproliferative disorders within 5 years (exceptions: basal cell carcinoma, localized squamous cell carcinoma, or cervical carcinoma in situ cured ≥1 year).
* Prosthetic joint infection (unless prosthesis removed/replaced ≥2 months before randomization).
* History of opportunistic infections (e.g., PJP, histoplasmosis, coccidioidomycosis).
* Active/latent TB infection (positive IGRA without clinical manifestations).
* Herpes infection:a) Active herpes zoster/simplex (HSV-1/2) at screening;b) History of severe herpes (disseminated disease, multidermatomal HSV, encephalitis, ophthalmic herpes, or recurrent zoster [≥2 episodes in 2 years]).
* History of severe bacterial, fungal, or viral infection requiring hospitalization for IV antibiotic or antiviral administration within 2 months before randomization.
* History of live vaccine administration within 2 months before randomization or plans to receive a live vaccine during the study period.
* Evidence of active infection and/or febrile illness requiring systemic anti-infective therapy within 2 weeks before randomization.
* Abnormal virology at screening:

  * HBsAg(+) or HBcAb(+) with detectable HBV-DNA
  * HCV Ab(+) with detectable HCV-RNA
  * History of HIV infection or HIV Ab(+)
  * Treponema pallidum Ab(+) with positive RPR/TRUST
* Prior use of TYK2 inhibitors (e.g., deucravacitinib).
* Use of any of the following therapeutic agents within 6 months before randomization:

  * IL-12/23, IL-17, or IL-23 inhibitors (ustekinumab, secukinumab, tildrakizumab, ixekizumab, guselkumab)
  * Rituximab or other B-cell depleting agents
  * Leflunomide
* Use of any of the following therapeutic agents within 3 months before randomization: Integrin pathway modulators (natalizumab) or B/T-cell modulators (alemtuzumab, abatacept, vedolizumab).
* Use of TNF inhibitors (etanercept, adalimumab, infliximab, certolizumab) within 2 months before randomization.
* Any biologic psoriasis therapy within 3 months or 5 half-lives (whichever longer) before randomization.
* Use of systemic non-biologic psoriasis agents and/or any systemic immunosuppressants within 4 weeks before randomization, including but not limited to: apremilast, methotrexate, azathioprine, cyclosporine, JAK inhibitors, 6-thioguanine, mercaptopurine, mycophenolate, hydroxyurea, tacrolimus, oral/injectable corticosteroids, retinoids, calcitriol/analogs, psoralen, sulfasalazine, fumarates).
* Use of Lithium, antimalarials, or intramuscular gold preparations within 4 weeks before randomization.
* Use of any botanical agents for the treatment of psoriasis or other immune disorders within 4 weeks before randomization, including herbal supplements or traditional Chinese medicines derived from plants, minerals, or animals.
* Received phototherapy within 4 weeks before randomization.
* Use of medicated shampoos and/or body washes within 2 weeks before randomization, including but not limited to products containing: corticosteroids, coal tar, >3% salicylic acid, vitamin D3 analogs.
* Use of any topical agents that may affect psoriasis symptoms within 2 weeks before randomization.
* Received any investigational therapy within 30 days or 5 half-lives (whichever is longer) before randomization, OR current participation in other trial.
* Laboratory values meeting any of the following criteria during screening or before randomization:

  * Liver: ALT/AST ≥3×ULN; total bilirubin >2×ULN
  * Hematology: WBC <3.0×10⁹/L (3000/mm³); ANC <1.0×10⁹/L (1000/mm³); lymphocyte count <0.5×10⁹/L (500/mm³); platelets <100×10⁹/L (100,000/mm³); hemoglobin <9.0 g/dL (90 g/L)
  * Renal: eGFR <60 mL/min/1.73m² (CKD-EPI equation)
* Pregnant or lactating women.
* Any condition deemed unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
Part 1：Incidence and Severity of Adverse Events (AEs) | 5 weeks
Part 2：Proportion of patients achieved Psoriasis Area Severity Index (PASI) 75 at Week 12 | Week 12
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity.
  PASI 75 is defined as the proportion of patients achieving ≥75% reduction in PASI score from baseline.

SECONDARY OUTCOMES:
Part 1： Changes from baseline in PASI | Week 4
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity.
Part 1： Changes from baseline in sPGA | Week 4
  Static Physician's Global Assessment (sPGA) is an average assessment of all psoriatic lesions, with scores ranging from 0 (indicating clear) to 5 (indicating severe).
Part 1： Changes from baseline in BSA | Week 4
  Body Surface Area (BSA) scores range from 0% (indicating absence of lesions) to 100% (indicating total body surface involvement), with higher scores correlating to greater disease severity.
Part 1： Changes from baseline in DLQI | Week 4
  Dermatology Life Quality Index（DLQI) total score ranges from 0 (indicating no impairment in quality of life) to 30 (indicating maximum impairment in quality of life).
Part 1：Proportion of patients achieving PASI 50/75/90/100 | Week 4
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity. PASI 50 is defined as the proportion of patients achieving ≥50% reduction in PASI score from baseline. PASI 75 is defined as the proportion of patients achieving ≥75% reduction in PASI score from baseline.PASI 90 is defined as the proportion of patients achieving ≥90% reduction in PASI score from baseline.PASI 100 is defined as the proportion of patients achieving ≥100% reduction in PASI score from baseline.
Part 2：Incidence and Severity of Adverse Events (AEs) | 16 weeks
Part 2：Proportion of patients achieving PASI 75 | Week 4 and 8
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity. PASI 75 is defined as the proportion of patients achieving ≥75% reduction in PASI score from baseline.
Part 2：Proportion of patients achieving PASI 50/90/100 | Week 4，8 and 12
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity. PASI 50 is defined as the proportion of patients achieving ≥50% reduction in PASI score from baseline. PASI 90 is defined as the proportion of patients achieving ≥90% reduction in PASI score from baseline.PASI 100 is defined as the proportion of patients achieving ≥100% reduction in PASI score from baseline.
Part 2：Proportion of patients achieving: (a) sPGA score of 0 or 1 with ≥2-point reduction from baseline (b) sPGA clearance (score 0) (c) Disease remission | Week 4，8 and 12
Part 2： Changes from baseline in PASI | Week 4，8 and 12
  Psoriasis Area and Severity Index (PASI) scores range from 0 to 72, with higher scores indicating more severe disease activity.
Part 2： Changes from baseline in BSA | Week 4，8 and 12
  Body Surface Area (BSA) scores range from 0% (indicating absence of lesions) to 100% (indicating total body surface involvement), with higher scores correlating to greater disease severity.
Part 2： Changes from baseline in sPGA | Week 4，8 and 12
  Static Physician's Global Assessment (sPGA) is an average assessment of all psoriatic lesions, with scores ranging from 0 (indicating clear) to 5 (indicating severe).
Part 2： Changes from baseline in DLQI | Week 4，8 and 12
  Dermatology Life Quality Index（DLQI) total score ranges from 0 (indicating no impairment in quality of life) to 30 (indicating maximum impairment in quality of life).
Pharmacokinetic parameters - Area Under the Curve(AUC) | Day 1~Day 85
Pharmacokinetic parameters - Peak Plasma Concentration (Cmax) | Day 1~Day 85

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Shiyan People's Hospital, Shiyan, Hubei
  - Shandong Provincial Hospital for Skin Diseases, Jinan, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University(Xibei Hospital ), Xi’an, Shanxi
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang
  - The First Affliated Hospital of Wenzhou Medical University, Wenzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: No